CLINICAL TRIAL: NCT06970353
Title: A Prospective, Single-Arm, Open-Label, Single-Center Phase II Exploratory Clinical Study to Evaluate the Efficacy and Safety of Tunlametinib in Subjects With NRAS-Mutant Locally Advanced or Metastatic Thyroid Cancer
Brief Title: Phase II Trial of Tunlametinib in NRAS-Mutant Advanced Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ji Dongmei, Associated Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-085-TC-002
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Radioactive Iodine-refractory, Differentiated Thyroid Cancer With NRAS Mutation; Advanced PDTC or ATC With NRAS Mutation
Keywords: NRAS mutant; Locally advanced thyroid cancer; Thyroid cancer; Metastatic thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Locally advanced or metastatic thyroid cancer with NRAS mutation (Experimental): Progressive locally advanced or metastatic radioactive iodine refractory NRAS mutant thyroid cancer
  Interventions: Drug: Tunlametinib; Drug: Tunlametinib+PD-1 mAb

INTERVENTIONS:
Drug: Tunlametinib — Locally advanced or metastatic radioactive iodine refractory NRAS mutant differentiated thyroid cancer
Drug: Tunlametinib+PD-1 mAb — Locally advanced or metastatic NRAS mutant poor-differentiated, undifferentiated thyroid cancer

SUMMARY:
This phase II trial evaluates Tunlametinib (MEK inhibitor) ± PD-1 in NRAS-mutant advanced thyroid cancer.

Key Objectives:

Assess efficacy (ORR by RECIST v1.1) Evaluate safety profiles

Study Design:

Single-arm, single-center 4 cohorts based on:

* Histology (differentiated vs. poorly/undifferentiated)
* Prior therapy status

Treatment:

* Cohorts 1-2: Tunlametinib monotherapy (12mg BID)
* Cohorts 3-4: Tunlametinib + PD-1 (commercially available)

Key Procedures:

Screening: NRAS testing + full staging (CT/MRI/PET) Monitoring: q3-week labs, q9-week imaging Follow-up: 30-day safety visit + q3-month survival tracking

Endpoints:

Primary: ORR Secondary: Safety (CTCAE), PFS, DoR

Unique Aspects:

First study targeting NRAS in thyroid cancer with MEK+PD-1 Includes rare aggressive subtypes (poorly/undifferentiated)

DETAILED DESCRIPTION:
Research Objective:

To evaluate the efficacy and safety of Tunlametinib (monotherapy or in combination with PD-1 mAb) in patients with locally advanced or metastatic NRAS-mutant thyroid cancer.

Study Endpoints:

Primary Endpoint:

Objective response rate (ORR) assessed per RECIST v1.1 (sum of partial and complete response rates).

Secondary Endpoints:

Efficacy:

Disease control rate (DCR) Duration of response (DoR) Time to response (TTR) Progression-free survival (PFS) Overall survival (OS), 6-month survival rate, 12-month survival rate

Safety:

Adverse events (AEs): Type, incidence, severity (graded by NCI-CTCAE v5.0), duration, and relationship to study treatment

Study Design:

This is a prospective, single-arm, open-label, single-center Phase II exploratory trial evaluating Tunlametinib ± PD-1 mAb in NRAS-mutant thyroid cancer.

Study Phases:

Screening: ≤28 days prior to enrollment (informed consent to baseline assessments).

Treatment: Until disease progression, intolerable toxicity, consent withdrawal, or investigator decision.

Follow-up:

Safety visit at 30 days (±7) post-treatment. Survival follow-up every 3 months (telephone/medical records).

Cohorts & Treatment:

Cohort 1 (n=10): Untreated, radioactive iodine-refractory, differentiated thyroid cancer.

Cohort 2 (n=10): Previously treated, radioactive iodine-refractory, differentiated thyroid cancer.

Regimen: Tunlametinib 12 mg BID (3-week cycles).

Cohort 3 (n=10): Untreated, poorly differentiated/anaplastic thyroid cancer.

Cohort 4 (n=10): Previously treated, poorly differentiated/anaplastic thyroid cancer.

Regimen: Tunlametinib 12 mg BID + PD-1 mAb(commercially available; per approved labeling).

Dose Adjustments:

Tunlametinib: Stepwise reduction (12 mg → 9 mg → 6 mg BID) for intolerance. Re-escalation permitted if toxicity resolves (e.g., 6 mg → 9 mg after ≥6 weeks).

PD-1: Adjusted per investigator judgment and drug labeling.

Efficacy Assessments:

Imaging (CT/MRI) every 9 weeks (3 cycles) per RECIST v1.1. Real-time ORR analysis by investigators and sponsor (Shanghai Kezhou Pharmaceutical).

Follow-up Procedures:

Safety visit: Day 30 (±7) post-treatment (vitals, labs, AE assessment). Survival follow-up: Quarterly until death/loss to follow-up/study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily join this study and sign an informed consent form;
2. Age: ≥ 18 years old, male or female not limited;
3. For locally advanced or recurrent/metastatic thyroid cancer diagnosed by histology and unable to undergo curative surgery, one of the following requirements must be met:

   1. Iodine refractory thyroid cancer;
   2. Differentiated thyroid cancer not suitable for iodine therapy;
   3. High grade, poorly differentiated or poorly differentiated thyroid cancer;
   4. Undifferentiated thyroid carcinoma;
4. Have undergone NGS testing (at our hospital or an external hospital), and be able to find that the test report or medical history has recorded a positive result for NRAS mutation in the gene test.
5. ECOG score 0-2 points; According to RECIST v1.1 evaluation, there is at least one assessable lesion;

7. Expected survival>12 weeks; 8. The main organ function and bone marrow function are normal.

* Blood routine: Hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); Absolute neutrophil count ≥ 1.5 × 109/L; platelet count ≥ 100 × 109/L;
* Liver function: Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) are ≤ 2.5 times the upper limit of normal (ULN). If there is liver metastasis, ALT and AST are ≤ 5 times ULN, and ALP is ≤ 6 times ULN; Total bilirubin ≤ 1.5 × ULN; Albumin ≥ 30 g/L;
* Renal function: serum creatinine ≤ 1.5 × ULN or creatinine clearance rate calculated by Cockroft Gault formula>60 mL/min;
* Cardiac function: Echocardiography shows a left ventricular ejection fraction (LVEF) of ≥ 55%; ECG QTcF ≤ 480ms; Creatine kinase (CK) ≤ 1 × ULN, troponin/hypersensitive troponin ≤ 1 × ULN;
* Coagulation function: International normalized ratio of prothrombin time (INR) ≤ 1.5 × ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; 9. Women of childbearing age must undergo a pregnancy test (serum or urine) with a negative result within 14 days before enrollment, and voluntarily use appropriate contraception methods during the observation period and within 3 months after the last administration of the study drug; For males, surgical sterilization or consent to use appropriate contraception methods during the observation period and within 3 months after the last administration of the study drug should be used.

Exclusion Criteria:

1. Within 4 weeks before the first medication, major surgery (excluding biopsy and outpatient minor surgery, such as placement of vascular access) or severe trauma occurred;
2. There are clinical symptoms of third interstitial fluid accumulation that cannot be controlled by drainage or other methods (such as a large amount of pleural fluid or ascites);
3. Cardiovascular and cerebrovascular diseases with impaired heart function or significant clinical significance, including but not limited to any of the following:

   Within 6 months prior to the start of treatment, acute coronary syndrome occurred, including acute myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, and stent implantation;
   * Symptomatic congestive heart failure (NYHA classification ≥ II); Evidence of clinically significant arrhythmia and/or conduction abnormalities within 6 months prior to the start of treatment or at present;
   * Poor control of hypertension (systolic blood pressure ≥ 140 and/or diastolic blood pressure ≥ 90 mmHg under medication control); Abnormal cardiac valve morphology (≥ grade 2) recorded by echocardiography, Note: Patients with grade 1 abnormal valve morphology (such as mild regurgitation/stenosis) are allowed to be enrolled, but patients with moderate valve thickening are prohibited from being enrolled;
   * History of congenital long QT syndrome; Or those who take drugs known to prolong the QT interval and cannot guarantee discontinuation during the study period;
4. Previous or screening retinal diseases, such as retinal vein occlusion (RVO), retinal artery occlusion, retinal vasculitis, diabetes retinopathy, hypertensive retinopathy, retinal telangiectasia (Costs disease), retinal pigment epithelial detachment (RPED), etc; Risk factors for RVO during screening (such as uncontrolled glaucoma or high intraocular pressure, history of high viscosity or hypercoagulability syndrome); Retinal diseases such as RPED;
5. Patients with interstitial lung disease or interstitial pneumonia, including clinically significant radiation pneumonitis (i.e. affecting daily living activities or requiring intervention treatment);
6. Positive for human immunodeficiency virus (HIV) antibodies, syphilis antibodies (Anti TP), hepatitis C virus (HCV) antibodies and HCV RNA, hepatitis B virus surface antigen (HBsAg) and HBV DNA (HBsAg positivity requires further testing for HBV DNA, HBV DNA ≥ 200 IU/ml, or ≥ 103 copies/ml);
7. History of allogeneic bone marrow transplantation or organ transplantation;
8. There are uncontrollable active infectious diseases (such as intravenous drip of antibiotics, antifungal or antiviral drugs) within 2 weeks before the first administration, or fever of unknown cause>38.5 ° C occurs during screening/before the first administration;
9. Irreversible electrolyte abnormalities (hypokalemia, hypomagnesemia, hypocalcemia detected by blood biochemistry);
10. Neuromuscular diseases related to CK elevation in the past or present (such as inflammatory myopathy, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy, rhabdomyolysis syndrome);
11. Arterial/venous thrombotic events that occur within 6 months prior to the first use of medication, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
12. Within 4 weeks prior to the first use of medication, the occurrence of Grade 3 bleeding symptoms as defined in the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0);
13. Patients with a history of other malignant tumors within the past 5 years, except for those who have been completely cured of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and cervical carcinoma in situ, and/or any malignant tumor patients who have been cured without disease or have had no disease for at least 5 consecutive years;
14. Individuals who are known to be allergic to any component of the investigational drug;
15. Have a clear history of neurological or mental disorders, including epilepsy and dementia;
16. Central nervous system (CNS) metastasis;
17. Prior to drug administration, all relevant anti-tumor treatment toxicity reactions (excluding hair loss, skin pigmentation, grade 1 chemotherapy related peripheral neurotoxicity, grade 2 toxicity caused by immune checkpoint inhibitors such as elevated blood glucose or hypothyroidism) did not recover to ≤ grade 1 levels (as determined by NCI CTCAE v5.0);
18. Uncontrolled concomitant diseases, including but not limited to severe diabetes (fasting blood glucose>250 mg/dl or 13.9 mmol/L), or other serious diseases requiring systemic treatment;
19. Vaccination with live or attenuated vaccine within 4 weeks prior to the first dose (note: if enrolled, subjects must not receive live vaccine during the study treatment period and within 30 days after the last dose of the study drug);
20. For premenopausal female subjects (postmenopausal female patients must have been menopausal for at least 12 months to be considered infertile), the pregnancy test result is positive; During the study period and at least 30 days after the last administration of the study drug, reproductive age subjects (including male subjects' reproductive age female spouses) who are expected to become pregnant, breastfeed, or unwilling to use effective contraceptive measures;
21. Patients who are known to be allergic to the components of the investigational drug or its analogues;
22. Patients who are receiving intravenous or oral medications that affect CYP isoenzymes (strong inducers and inhibitors of CYP2C9 and CYP3A4) and cannot discontinue the protocol at least one week before starting study treatment and during the study period; I am currently taking drugs with a narrow therapeutic window that are metabolized by CYP1A2;
23. Inability to swallow capsules or intractable nausea and vomiting, malabsorption, extracorporeal bile diversion, or any significant small bowel resection that may hinder the full absorption of the study drug;
24. Other situations that researchers consider unsuitable for inclusion. If accompanied by family or social factors, it may affect the safety of the subjects or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to approximately 3-5 years
  Complete remission rate and partial remission rate

SECONDARY OUTCOMES:
Disease Control Rate | up to approximately 3-5 years
  Complete remission rate and partial remission rate and stable disease rate
Duration of Response | up to approximately 3-5 years
  Time from the date of first partial remission or complete remission to the date of disease progression, or death of any cause, or date of lost follow-up, whichever comes first, otherwise subject data were censored at time last known disease free.
Time to Response | up to approximately 3-5 years
  Time from the initiation of the treatment to the first remission
Progression-free Survival | up to approximately 3-5 years
  Time from the date of enrollment to of disease progression, or death of any cause, or date of lost follow-up, whichever comes first, otherwise subject data were censored at time last known disease free.
Overall Survival | up to approximately 3-5 years
  Time from the date of enrollment to data of death from any cause, or date of lost follow-up, whichever comes first, and otherwise censored at time last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Long Wang, M.D, Principal Investigator — Fudan University; Qing-Hai Ji, M.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No